CLINICAL TRIAL: NCT01129583
Title: Intraoperative Injection of Botulinum Toxin A (Botox) for the Prevention of Post-Traumatic Elbow Stiffness: A Randomized Double Blind Placebo Controlled Study
Brief Title: Botulinum Toxin as a Novel Treatment for Prevention of Post-Traumatic Elbow Stiffness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Melvin Rosenwasser, Robert E. Carroll Professor of Surgery of the Hand in the Department of Orthopaedic Surgery at the New York-Presbyterian Hospital at the Columbia University Medical Center, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AAAA8392
Record Dates: First submitted 2010-05-21; First posted 2010-05-24 (Estimated); Results first posted 2011-05-02 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Post Traumatic Stiffness
Keywords: Botulinum Toxin; Elbow Stiffness
MeSH Terms: interventions — Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botulinum Toxin (Experimental): 100 U injected into biceps, 100 U into brachialis
  Interventions: Drug: Botulinum Toxin Type A
- Saline (Placebo Comparator): 100 U injected into biceps, 100 U into brachialis
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Botulinum Toxin Type A — Injection into the biceps brachii and brachialis immediately following the initial fracture surgery
  Other Names: Botox®
  Arms: Botulinum Toxin
Drug: Saline — Injection into the biceps brachii and brachialis immediately following the initial fracture surgery
  Arms: Saline

SUMMARY:
This is a randomized double blind placebo controlled study to investigate the hypothesis that injection of botulinum toxin A into the muscles surrounding the elbow following the surgical treatment of an elbow fracture will reduce postoperative stiffness and improve function.

DETAILED DESCRIPTION:
This is a randomized double blind placebo controlled prospective study in which botulinum toxin A (Botox®) or normal saline will be intraoperatively injected into the muscles surrounding the elbow following the surgical treatment of an elbow fracture or elbow fracture dislocation.

Eligible patients will be identified by the Principal Investigator in his practice or by fellows and residents from the clinic population and emergency department admissions. After providing informed consent, all subjects will undergo a baseline examination that will include a medical and orthopaedic history, physical examination, and radiographs. The surgical procedure itself will not differ from the standard care for elbow fractures. The only difference is injection of Botox® or normal saline into the muscles of the injured arm. Subjects will undergo post-operative evaluation at various intervals for up to two years. The study and control group will be compared to each other and to contralateral arms in regards to elbow range of motion, patient questionnaire scores (DASH) and an observer-based elbow scoring system (Broberg and Morrey).

Traumatic injury to the elbow resulting in a fracture or fracture/dislocation of the elbow often leads to a stiff elbow with limited function. Posttraumatic elbow stiffness is a common problem that is difficult to manage. The best way to decrease the morbidity is through prevention. An intraoperative injection of Botox® has been effective in treating upper limb spasticity disorders and may prevent the development of elbow stiffness, and decrease the need for future surgery to regain motion.

ELIGIBILITY:
Inclusion Criteria:

* Capable of providing informed consent
* 18 years old and older
* Elbow fractures that require operative intervention including:
* Supracondylar distal humerus fractures
* Intra-articular distal humerus fractures
* Proximal ulna and radius fractures

Exclusion Criteria:

* Patients less than 18 years old
* Injuries that do not normally require surgical repair
* Patients with underlying spasticity
* Patients with burns about the elbow
* Patients with extensive soft tissue injuries of the elbow
* Patients with head or spinal cord injuries
* Myasthenia gravis, Eaton-Lambert, amyotrophic lateral sclerosis or any other disease that interferes with neuromuscular function
* Use of aminoglycoside antibiotics or other drug therapies that interfere with neuromuscular function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2003-11; Primary Completion 2009-09 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melvin Rosenwasser, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the orthopaedic upper extremity trauma clinic of the primary investigator. The recruitment period was 49 months in length, from 11/2003 through 11/2007.
Pre-assignment Details: Of the 59 patients assessed for eligibility, 41 patients were excluded based on the listed inclusion/exclusion criteria.
Groups:
- Botulinum Toxin; Saline: Intraoperative injection of 100 U into biceps and 100 U into brachialis following surgical treatment of an elbow fracture or elbow fracture dislocation.
Period: Overall Study
Arm/Group | Botulinum Toxin | Saline
Started | 9 | 9
Completed | 6 | 7
Not Completed | 3 | 2
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Ipsilateral Upper Extremity Injury | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Botulinum Toxin | Saline | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 16
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (13) | 45 (21) | 49 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 6 | 5 | 11
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Disabilities of the Arm, Shoulder, and Hand (DASH) Questionnaire
Description: The Disabilities of the Arm, Shoulder and Hand (DASH) Outcome Measure is a questionnaire designed to measure physical function and symptoms in patients with musculoskeletal disorders of the upper limb.
  The DASH is scored in two components: the disability/symptom questions (30 items, scored 1-5) and the optional high performance sport/music or work section (4 items, scored 1-5). The DASH disability/symptom score (0-100) is calculated by averaging all the scores, subtracting one and multiplying by 25. A score of 0 represents "no disability", while 100 represents "maximum possible disability".
Time Frame: 1 year post-op
Measure: Mean (Standard Error); unit: Scores on a Scale (0-100)
Arm/Group | Botulinum Toxin | Saline
Number analyzed (Participants) | 9 | 9
Scores on a Scale (0-100) | 27 (11) | 54 (8)
Statistical Analysis 1: Comparison: Botulinum Toxin vs Saline; Test type: Superiority or Other; p = 0.06, t-test, 2 sided

2. Secondary Outcome: Elbow Range of Motion
Description: Elbow flexion/extension active range of motion was assessed with the use of a standard goniometer with the center placed over the lateral epicondyle and the arms aligned with the long axis of the humerus and ulna, respectively. Full extension (arm completely straight) is defined as 0 degrees, and peak flexion is measured as the angle formed by the arm and forearm compared to a full straight arm.
Time Frame: 3 months post-op
Measure: Mean (Standard Error); unit: Degrees
Arm/Group | Botulinum Toxin | Saline
Number analyzed (Participants) | 9 | 9
Degrees | 103 (7.6) | 73 (6.3)
Statistical Analysis 1: Comparison: Botulinum Toxin vs Saline; Test type: Superiority or Other; p = 0.01, t-test, 2 sided

3. Secondary Outcome: Broberg Morrey Composite Elbow Function Score
Description: Composite elbow function store that takes into account range of motion, stability, strength, and pain. Score ranges from 0 (worse possible function) to 100 (best possible function).
Time Frame: 6 months post-op
Measure: Mean (Standard Error); unit: Score
Arm/Group | Botulinum Toxin | Saline
Number analyzed (Participants) | 9 | 9
Score | 82 (1.9) | 65 (2.9)
Statistical Analysis 1: Comparison: Botulinum Toxin vs Saline; Test type: Superiority or Other; p = 0.02, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Botulinum Toxin | Saline
Serious Adverse Events (participants affected / at risk) | 1/9 | 0/9
Other Adverse Events (participants affected / at risk) | 1/9 | 1/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Botulinum Toxin (N=9) | Saline (N=9)
Death (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Botulinum Toxin (N=9) | Saline (N=9)
Unrelated Upper Extremity Injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
* Limited statistical power: Limitations in time and funding as well as difficulties in recruiting
* Blinding challenges: Weakness in the flexor muscles of patients receiving botulinum toxin injections was clinically apparent

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No